CLINICAL TRIAL: NCT03504709
Title: Advanced MRI and EEG to Predict Recovery of Consciousness After Severe Traumatic Brain Injury
Brief Title: REsting and Stimulus-based Paradigms to Detect Organized NetworkS and Predict Emergence of Consciousness
Acronym: RESPONSE 2
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Brian L. Edlow, M.D., Neurocritical Care Faculty, Massachusetts General Hospital, Associate Director, Center for Neurotechnology and Neurorecovery (CNTR) Director, Laboratory for NeuroImaging of Coma and Consciousness (NICC), Massachusetts General Hospital
Other Study IDs: 2012P000784
Record Dates: First submitted 2018-03-20; First posted 2018-04-20 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Consciousness Disorder; Coma; Brain Injuries, Traumatic
MeSH Terms: conditions — Consciousness Disorders; Coma; Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient (n=50): Adults with acute severe traumatic brain injury who undergo advanced neuroimaging and electrophysiological studies while in the intensive care unit and are followed for 6 months post injury.
- Healthy (n=25): Healthy adults with no neurological, psychiatric, or medical disease.

SUMMARY:
The aim of this study is to assess the utility of advanced magnetic resonance imaging (MRI) and electroencephalographic (EEG) technologies for predicting functional outcomes in patients with severe traumatic brain injury (TBI).

ELIGIBILITY:
Patients:

Inclusion Criteria:

* Traumatic Brain Injury
* Glasgow Coma Scale score of 3-8 within 24 hours, unconfounded by sedation, paralysis, hypoxia, hypotension, hypothermia, or concurrent medical illness
* Clinical evidence of disorder of consciousness defined as coma, VS, or MCS

Exclusion Criteria:

* History of prior severe brain injury or dementia
* Emergence from MCS at time of initial CRS-R assessment

Healthy Subjects:

Exclusion Criteria:

History of brain injury or neurological disease, psychiatric disease, or any history of diabetes, high blood pressure, heart disease, or kidney disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults admitted to the intensive care unit for acute severe traumatic brain injury
Sampling Method: Non-Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2018-09-05 (Actual); Primary Completion 2023-07-19 (Actual); Study Completion 2023-10-23 (Actual)

PRIMARY OUTCOMES:
Disability Rating Scale total score | 6 months post injury
  The Disability Rating Scale (DRS) provides quantitative information regarding functional disability in patients recovering from severe brain injury. The total score on the DRS ranges from 0 to 29 with higher scores indicating a greater degree of disability. DRS subscale scores include eye opening [score range 0-3], communication [score range 0-4], motor response [score range 0-5], cognitive ability for feeding [score range 0-3], cognitive ability for toileting [score range 0-3], cognitive ability for grooming [score range 0-3], level of function [score range 0-5], and employability [score range 0-3]. Subscale scores are summed to produce the total score.

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Edlow BL, Chatelle C, Spencer CA, Chu CJ, Bodien YG, O'Connor KL, Hirschberg RE, Hochberg LR, Giacino JT, Rosenthal ES, Wu O. Early detection of consciousness in patients with acute severe traumatic brain injury. Brain. 2017 Sep 1;140(9):2399-2414. doi: 10.1093/brain/awx176. PMID 29050383
- [Background] Bodien YG, Giacino JT, Edlow BL. Functional MRI Motor Imagery Tasks to Detect Command Following in Traumatic Disorders of Consciousness. Front Neurol. 2017 Dec 18;8:688. doi: 10.3389/fneur.2017.00688. eCollection 2017. PMID 29326648
- [Background] Bodien YG, Chatelle C, Edlow BL. Functional Networks in Disorders of Consciousness. Semin Neurol. 2017 Oct;37(5):485-502. doi: 10.1055/s-0037-1607310. Epub 2017 Dec 5. PMID 29207410
- [Background] Threlkeld ZD, Bodien YG, Rosenthal ES, Giacino JT, Nieto-Castanon A, Wu O, Whitfield-Gabrieli S, Edlow BL. Functional networks reemerge during recovery of consciousness after acute severe traumatic brain injury. Cortex. 2018 Sep;106:299-308. doi: 10.1016/j.cortex.2018.05.004. Epub 2018 May 12. PMID 29871771
- [Derived] Olchanyi MD, Augustinack J, Haynes RL, Lewis LD, Cicero N, Li J, Destrieux C, Folkerth RD, Kinney HC, Fischl B, Brown EN, Iglesias JE, Edlow BL. Automated MRI Segmentation of Brainstem Nuclei Critical to Consciousness. Hum Brain Mapp. 2025 Oct 1;46(14):e70357. doi: 10.1002/hbm.70357. PMID 41074651